CLINICAL TRIAL: NCT02808715
Title: Identification and Metabolic Characterization of a Cohort of Human Subjects With Mutations in PRDM-16
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/337/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Mutation; Obesity; Dyslipidemia; Diabetes
MeSH Terms: conditions — Obesity; Dyslipidemias; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample will be obtained and processed to isolate genomic DNA. A PCR-based strategy will be employed to sequence the entire PRDM-16 locus to identify variants. Variant alleles of PRDM-16 will be classified as having benign or deleterious mutations. Subjects who harbor deleterious mutations in both alleles of PRDM-16 will be identified for further study.
  For subjects who withdraw from the study, no further testing of the blood samples will occur. The blood will be stored at the NHRIS biobank. After the study is complete the samples will remain in storage at the NHRIS biobank.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood Sample Collection — Blood draw #1 Site of blood draw: IMU Volume of blood: 20mL Purpose of blood draw: Isolation of genomic DNA Site of storage: NHRIS biobank Coding: Specimens will be identified using a research ID that will be affixed to samples using bar-coding. After the blood is collected, stored the blood at 4 degree Celsius and contact the NHCS biobank coordinator to collect the blood samples. The blood samples must be collected within 1 hour of collection.

SUMMARY:
Chinese male subjects will be invited to participate in a research study of brown fat, a special tissue in the body that is designed to burn energy to make heat. The objective is to learn the importance of a gene called "PRDM-16" for the function of brown fat. Subjects were selected as a possible subject in this study because they fulfil the age and weight criteria.

500 subjects from the Singhealth Investigational Medicine Unit healthy volunteer database will be recruited over a period of 2 years. All of the subjects will have their PRDM-16 gene sequenced. The objective is to identify subjects with mutations, or changes, in their PRDM-16 gene. About 12 subjects with PRDM-16 mutations are expected to be identified.

Samples of blood obtained during the course of this study will be stored and analysed only for the purposes of this study for a period not exceeding 2 years, and will be destroyed after completion of the study, unless subject is agreeable to donate the samples to the National Heart Centre Singapore for continuous storage for future studies that are approved by the institutional review board..

DETAILED DESCRIPTION:
The long-term objective of this study is to develop new treatments for obesity and obesity-associated disorders such as diabetes and dyslipidemia. The recent finding of active brown fat depots in adult humans provides an exciting new strategy for the treatment of these diseases. Brown fat is a specialized organ found primarily in small mammals. Brown fat has the unique capability to burn fuel at high rates in order to generate heat. The role of brown fat in mammals is to defend against cold exposure. Human infants have active brown fat deposits located in the intra-scapular region. This brown fat depot regresses with age and it was long thought that adult humans had no brown fat tissue. Recent studies have demonstrated the presence of brown fat activity in adult humans following exposure to cold. Brown fat in adult humans is concentrated in the cervical region and displays some sex-specific differences. Furthermore the size of the depot is inversely correlated with BMI and age of the subjects. This finding has generated intense interest as it opens up the possibility of harnessing brown fat as a means of combating obesity and obesity-related disorders in man. Indeed, maneuvers that activate brown fat in humans have been shown to cause reductions in fat mass.

Much of our understanding of brown fat biology comes from work in mice. Of particular relevance for the treatment of human disease are several findings. First, increasing brown fat activity in mice renders the animals resistant to the development of obesity on a high fat diet. Second, levels of insulin sensitivity are directly related to brown fat activity. Finally, the transcription factor factor PR-domain containing protein 16 (PRDM-16) is crucial for directing the biology of brown fat.

The overall goal of the study is to translate the findings from mouse studies of brown fat into human subjects. This is an important first step in the process of developing brown fat-targeted therapies to treat human metabolic diseases such as obesity and insulin resistance. In view of this the investigators are interested in answering several questions. First, do humans with mutations in PRDM-16 have defects in brown fat activity? Recently, humans with mutations in PRDM-16 were identified and found to have a cardiomyopathy phenotype. The brown fat function in these individuals has not been described. By employing a genetic screen of volunteers the investigators hope to identify subjects in Singapore with defects in PRDM-16. Prior studies in humans suggest that the size of the brown fat depot is inversely correlated with BMI and age of the subjects and that depot size varies between the sexes. In order to eliminate BMI, age and sex as confounding variables the investigators will include male subjects of Chinese race between the ages of 21 and 50 and with BMI greater than 18.5 but less than 30. The investigators will include only Chinese subjects to avoid confounding our initial study with variables that relate to race of the subjects. The identification of human subjects carrying mutations in PRDM-16 will set the stage for further studies that will attempt to several research questions. These include whether humans with PRDM-16 mutations have defects in brown fat and the metabolic consequences for humans with defective brown fat.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese
* Age >= 21 and =< 50
* BMI >=18.5 and =< 30
* Ability to provide written, informed consent.
* To control for this the investigators will include only adult Chinese men less than 50 years old.
* Since obesity also alters brown fat function the investigators will exclude those with BMI>30.

Exclusion Criteria:

* Diagnosis of DM2
* Use of beta blockers, TZD (ie rosiglitazone/pioglitazone) or metformin Since the subjects will be recruited from the IMU healthy volunteer database there should be no prior history of DM2 or medication use. Nevertheless, diagnosis of DM2 and use of the drugs listed can alter brown fat activity and interfere with our analysis.
* Presence of pacemakers or foreign metallic objects in the eyes. Future planned experiments with the identified cohort include cardiac MRI. Subjects with pacemakers or foreign metallic objects in the eyes will be ineligible for this potential follow-up study.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 500 subjects will be recruited from the IMU healthy volunteer database. The investigators will enroll male Chinese volunteers. Women, children and the elderly are excluded from our initial study since prior research suggests that age and sex has an effect on brown fat function. In order to study the role of PRDM-16 in brown fat function the investigators wish to keep other contributing variables static in our study.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with deleterious mutations in the PRDM-16 locus, using standard genomic methods | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tan Ru San, MBBS, Principal Investigator — National Heart Centre Singapore

IPD SHARING:
Plan to Share IPD: No